CLINICAL TRIAL: NCT01022957
Title: Characterization and Analysis of Long-term Evolution of Renal and Extra-renal Damages in the Course of Nephronophthisis
Brief Title: Nephronophthisis : Clinical and Genetic Study
Acronym: NEPHAER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P050605
Record Dates: First submitted 2009-11-30; First posted 2009-12-01 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Nephronophthisis
Keywords: extra renal damages
MeSH Terms: conditions — Nephronophthisis, familial juvenile

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Study group (Experimental): Neurological, ophthalmological, olfactive exams and cerebral MRI
  Interventions: Genetic: genetic diagnosis

INTERVENTIONS:
Genetic: genetic diagnosis — to determine the long term evolution of Nephronophthisis in terms of renal disease as well as extra-renal damages for patients having a confirmed diagnosis of NPHP1, NPHP2, NPHP3, NPHP4, NPHP5, NPHP6 or NPHP8 gene mutation

SUMMARY:
to describe evolution of Nephronophthisis

DETAILED DESCRIPTION:
To specify the long term evolution of Nephronophthisis in terms of renal disease as well as extra-renal damages for patients having a confirmed diagnosis of NPHP1, NPHP2, NPHP3, NPHP4, NPHP5, NPHP6 or NPHP8 gene mutation

ELIGIBILITY:
Inclusion Criteria:

* NPHP1, NPHP2, NPHP3, NPHP4, NPHP5, NPHP6 or NPHP8 gene mutation
* 7 years old and older

Exclusion Criteria:

* MRI contra-indications

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2006-11; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
to determine the long term evolution of Nephronophthisis in terms of renal disease as well as extra-renal damages for patients having a confirmed diagnosis of NPHP1, NPHP2, NPHP3, NPHP4, NPHP5, NPHP6 or NPHP8 gene mutation | start from the first time of clinical diagnosis to now

SECONDARY OUTCOMES:
to study siblings to anticipate clinical complications (renal and extra-renal damages) of Nephronophthisis

CONTACTS AND LOCATIONS:
Overall Officials: Rémi SALOMON, MD, PhD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hopital Necker, Paris, France